CLINICAL TRIAL: NCT00846859
Title: Does Varenicline Influence Alcohol Consumption in Alcohol Dependent Individuals?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Karolinska University Hospital (Other); Malmö University (Other)
Responsible Party: Bo Söderpalm/ MD, PhD, sponsor, Addiction Biology Unit, Sahlgrenska University Hospital, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GOTABU-BO2
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Alcohol Dependence
Keywords: alcohol dependence; nicotine dependence; alcohol abuse; varenicline; Champix; Chantix; smoking; drinking; snuffing; diary; phosphatidyl ethanol; PEth
MeSH Terms: conditions — Alcoholism; Tobacco Use Disorder; Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- varenicline (Experimental)
  Interventions: Drug: varenicline (Champix/Chantix)
- placebo (Placebo Comparator)
  Interventions: Drug: placebo for varenicline

INTERVENTIONS:
Drug: varenicline (Champix/Chantix) — 14 weeks of per oral tablet treatment in an escalating dosing regimen (0.5 mg - 1.0 mg/day; 1 - 2 tablets/day).
  Other Names: Champix(R)/Chantix(R)
  Arms: varenicline
Drug: placebo for varenicline — 14 weeks of per oral tablet treatment in an escalating dosing regimen (1 - 2 tablets/day)
  Other Names: placebo for Champix(R) / Chantix(R)
  Arms: placebo

SUMMARY:
The aim of the present clinical trial is to investigate whether 14 weeks of treatment with a prescription medication for smoking cessation (European trade name: Champix(R); US trade name: Chantix(R)), can reduce alcohol consumption in alcohol dependent individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 30-70 years at screening
2. Alcohol dependence according to DSM-IV (meeting ≥3 out of 7 criteria)
3. ≥ 20 heavy drinking days (men: ≥ 5 drinks/day, women: ≥4 drinks/day, where 1 std. drink is defined as 12 g ethanol) during the last 60 days
4. Participants must have signed the informed consent

Exclusion Criteria:

1. Subject to treatment of alcohol withdrawal within 30 days of study initiation
2. Subject to treatment that may affect alcohol consumption including acamprosate, naltrexone, disulfiram, ondansetron, topiramate, SSRIs, varenicline, mirtazapine, rimonabant, methylphenidate or atomoxetine within 3 months of study initiation
3. Subject to treatment of depression within 3 months of study initiation
4. The continuous use of drugs such as codeine, hydroxyzine, alimemazine, benzodiazepines or sedatives (the sporadic use of these compounds is accepted)
5. Any concurrent medication that may affect the results of the trial or is considered to compromise the safety of the participants in the trial
6. History of Delirium Tremens the last 5 years or any history of abstinence-induced seizures
7. Laboratory hepatic values of more than 3 times the upper limit of the normal range or other clinically significant abnormalities in the screening laboratory values.
8. Participants who are pregnant or nursing infant(s), and women of childbearing potential not using a contraceptive method judged by the investigator to be effective.
9. Any ongoing serious psychiatric or somatic disorder
10. Any psychiatric Axel I diagnoses (except for nicotine or alcohol dependence)
11. The concurrent use of illicit drugs based on urine-toxicity test
12. The need for detoxification
13. Diabetes Mellitus Type 1
14. Suicidal risk
15. Homelessness
16. Additional factors that implies to the investigator/physician that the participant will not be completing the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption as measured by diary and questionnaires: the number of heavy drinking days (as percentage) defined as ≥5 standard drinks per day for men and ≥4 standard drinks per day for women

SECONDARY OUTCOMES:
Alcohol consumption as measured by diary and questionnaires: total amount (grams) of consumed alcohol compared to baseline.
Percentage (and number) of abstaining days compared to baseline.
Drinks per drinking day compared to baseline.
Alcohol consumption as measured by alcohol markers in blood compared to baseline.
Nicotine use in alcohol dependent subjects as measured by diary and questionnaires compared to baseline.
Compliance as measured by diary and returned medication packages.

CONTACTS AND LOCATIONS:
Overall Officials: Elin Löf, PhD, Study Director — Addiction Biology Unit, University of Gothenburg and Beroendekliniken, Sahlgrenska University Hospital, Sweden; Bo Söderpalm, MD, PhD, Principal Investigator — Addiction Biology Unit, University of Gothenburg and Beroendekliniken, Sahlgrenska University Hospital, Sweden
Locations (3):
- Sweden (3):
  - Addiction Biology Unit, Beroendekliniken, University of Gothenburg and Sahlgrenska University Hospital, Gothenburg
  - Beroendecentrum, Malmö University Hospital (UMAS), Sweden, Malmo
  - Department of Clinical Neuroscience Section of Dependence Research Magnus Huss Clinic: M4:02 Karolinska University Hospital, Stockholm

REFERENCES:
- [Background] Ericson M, Lof E, Stomberg R, Soderpalm B. The smoking cessation medication varenicline attenuates alcohol and nicotine interactions in the rat mesolimbic dopamine system. J Pharmacol Exp Ther. 2009 Apr;329(1):225-30. doi: 10.1124/jpet.108.147058. Epub 2009 Jan 6. PMID 19126781
- [Background] Lof E, Olausson P, deBejczy A, Stomberg R, McIntosh JM, Taylor JR, Soderpalm B. Nicotinic acetylcholine receptors in the ventral tegmental area mediate the dopamine activating and reinforcing properties of ethanol cues. Psychopharmacology (Berl). 2007 Dec;195(3):333-43. doi: 10.1007/s00213-007-0899-4. Epub 2007 Aug 17. PMID 17703283
- [Background] Lof E, Chau PP, Stomberg R, Soderpalm B. Ethanol-induced dopamine elevation in the rat--modulatory effects by subchronic treatment with nicotinic drugs. Eur J Pharmacol. 2007 Jan 26;555(2-3):139-47. doi: 10.1016/j.ejphar.2006.10.056. Epub 2006 Oct 28. PMID 17141214
- [Background] Soderpalm B, Ericson M, Olausson P, Blomqvist O, Engel JA. Nicotinic mechanisms involved in the dopamine activating and reinforcing properties of ethanol. Behav Brain Res. 2000 Aug;113(1-2):85-96. doi: 10.1016/s0166-4328(00)00203-5. PMID 10942035
- [Background] Ericson M, Blomqvist O, Engel JA, Soderpalm B. Voluntary ethanol intake in the rat and the associated accumbal dopamine overflow are blocked by ventral tegmental mecamylamine. Eur J Pharmacol. 1998 Oct 9;358(3):189-96. doi: 10.1016/s0014-2999(98)00602-5. PMID 9822883
- [Background] Blomqvist O, Ericson M, Engel JA, Soderpalm B. Accumbal dopamine overflow after ethanol: localization of the antagonizing effect of mecamylamine. Eur J Pharmacol. 1997 Sep 10;334(2-3):149-56. doi: 10.1016/s0014-2999(97)01220-x. PMID 9369343
- [Background] Blomqvist O, Soderpalm B, Engel JA. Ethanol-induced locomotor activity: involvement of central nicotinic acetylcholine receptors? Brain Res Bull. 1992 Aug;29(2):173-8. doi: 10.1016/0361-9230(92)90023-q. PMID 1525672
- [Background] Blomqvist O, Engel JA, Nissbrandt H, Soderpalm B. The mesolimbic dopamine-activating properties of ethanol are antagonized by mecamylamine. Eur J Pharmacol. 1993 Nov 9;249(2):207-13. doi: 10.1016/0014-2999(93)90434-j. PMID 8287902
- [Background] Steensland P, Simms JA, Holgate J, Richards JK, Bartlett SE. Varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, selectively decreases ethanol consumption and seeking. Proc Natl Acad Sci U S A. 2007 Jul 24;104(30):12518-23. doi: 10.1073/pnas.0705368104. Epub 2007 Jul 11. PMID 17626178
- [Background] Blomqvist O, Hernandez-Avila CA, Van Kirk J, Rose JE, Kranzler HR. Mecamylamine modifies the pharmacokinetics and reinforcing effects of alcohol. Alcohol Clin Exp Res. 2002 Mar;26(3):326-31. PMID 11923584
- [Background] Young EM, Mahler S, Chi H, de Wit H. Mecamylamine and ethanol preference in healthy volunteers. Alcohol Clin Exp Res. 2005 Jan;29(1):58-65. doi: 10.1097/01.alc.0000150007.34702.16. PMID 15654292
- [Background] Chi H, de Wit H. Mecamylamine attenuates the subjective stimulant-like effects of alcohol in social drinkers. Alcohol Clin Exp Res. 2003 May;27(5):780-6. doi: 10.1097/01.ALC.0000065435.12068.24. PMID 12766622
- [Background] Rollema H, Chambers LK, Coe JW, Glowa J, Hurst RS, Lebel LA, Lu Y, Mansbach RS, Mather RJ, Rovetti CC, Sands SB, Schaeffer E, Schulz DW, Tingley FD 3rd, Williams KE. Pharmacological profile of the alpha4beta2 nicotinic acetylcholine receptor partial agonist varenicline, an effective smoking cessation aid. Neuropharmacology. 2007 Mar;52(3):985-94. doi: 10.1016/j.neuropharm.2006.10.016. Epub 2006 Dec 8. PMID 17157884
- [Background] Tonstad S. Varenicline for smoking cessation. Expert Rev Neurother. 2007 Feb;7(2):121-7. doi: 10.1586/14737175.7.2.121. PMID 17286546
- [Background] Jorenby DE, Hays JT, Rigotti NA, Azoulay S, Watsky EJ, Williams KE, Billing CB, Gong J, Reeves KR; Varenicline Phase 3 Study Group. Efficacy of varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs placebo or sustained-release bupropion for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):56-63. doi: 10.1001/jama.296.1.56. PMID 16820547
- [Background] Gonzales D, Rennard SI, Jorenby DE, Reeves KR. Comment: Oral varenicline for smoking cessation. Ann Pharmacother. 2007 Apr;41(4):720-1. doi: 10.1345/aph.1H310a. Epub 2007 Mar 20. No abstract available. PMID 17374627
- [Background] Daeppen JB, Smith TL, Danko GP, Gordon L, Landi NA, Nurnberger JI Jr, Bucholz KK, Raimo E, Schuckit MA. Clinical correlates of cigarette smoking and nicotine dependence in alcohol-dependent men and women. The Collaborative Study Group on the Genetics of Alcoholism. Alcohol Alcohol. 2000 Mar-Apr;35(2):171-5. doi: 10.1093/alcalc/35.2.171. PMID 10787393
- [Background] Larsson A, Jerlhag E, Svensson L, Soderpalm B, Engel JA. Is an alpha-conotoxin MII-sensitive mechanism involved in the neurochemical, stimulatory, and rewarding effects of ethanol? Alcohol. 2004 Oct-Nov;34(2-3):239-50. doi: 10.1016/j.alcohol.2004.10.002. PMID 15902919
- [Background] Larsson A, Svensson L, Soderpalm B, Engel JA. Role of different nicotinic acetylcholine receptors in mediating behavioral and neurochemical effects of ethanol in mice. Alcohol. 2002 Nov;28(3):157-67. doi: 10.1016/s0741-8329(02)00244-6. PMID 12551757
- [Background] Larsson A, Edstrom L, Svensson L, Soderpalm B, Engel JA. Voluntary ethanol intake increases extracellular acetylcholine levels in the ventral tegmental area in the rat. Alcohol Alcohol. 2005 Sep-Oct;40(5):349-58. doi: 10.1093/alcalc/agh180. Epub 2005 Jul 25. PMID 16043436
- [Background] Bohn MJ, Babor TF, Kranzler HR. The Alcohol Use Disorders Identification Test (AUDIT): validation of a screening instrument for use in medical settings. J Stud Alcohol. 1995 Jul;56(4):423-32. doi: 10.15288/jsa.1995.56.423. PMID 7674678
- [Background] Anton RF, Moak DH, Latham P. The Obsessive Compulsive Drinking Scale: a self-rated instrument for the quantification of thoughts about alcohol and drinking behavior. Alcohol Clin Exp Res. 1995 Feb;19(1):92-9. doi: 10.1111/j.1530-0277.1995.tb01475.x. PMID 7771669
- [Background] Wilson CB, Gutin P, Boldrey EB, Drafts D, Levin VA, Enot KJ. Single-agent chemotherapy of brain tumors. A five-year review. Arch Neurol. 1976 Nov;33(11):739-44. doi: 10.1001/archneur.1976.00500110007002. PMID 185991